CLINICAL TRIAL: NCT01842191
Title: Efficacy of Fish Oil on Serum TNFα, IL-1β, IL-6, Oxidative Stress Markers in Multiple Sclerosis Treated With Interferon Beta 1-b
Brief Title: Efficacy of Fish Oil in Multiple Sclerosis
Acronym: EFOMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Genaro Gabriel Ortiz, Investigador titular D, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FOMS
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Relapsing- Remitting Multiple Sclerosis
Keywords: R-R MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fish Oils; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Experimental)
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil — Patients received 4g/day Omega Rx capsules (Dr. Sears zone diet) containing 0.8 g EPA and 1.6 g DHA and excipient (glycerin, water purified, tocopherol, sunflower oil and titanium dioxide), during 12 months.
  Other Names: PUFAS; Omega 3
  Arms: Fish oil
Dietary Supplement: Placebo — Orally, 4 Capsules per day, (glycerin, water purified, tocopherol, sunflower oil and titanium dioxide), during 12 months.
  Other Names: Control
  Arms: Placebo

SUMMARY:
The aim of the present work was to evaluate the efficacy of fish oil supplementation on serum proinflammatory cytokines levels, oxidative stress markers and disease progression in MS.

DETAILED DESCRIPTION:
Current research findings suggest that Omega-3 polyunsaturated fatty acids (PUFA) such as eicosahexanoic acid (EPA) and docosahexaenoic acid (DHA) contained in fish oil may have anti-inflammatory, antioxidant and neuroprotective effects. The aim of the present work was to evaluate the efficacy of fish oil supplementation on serum proinflammatory cytokines levels, oxidative stress markers and disease progression in MS. 50 patients with relapsing-remitting MS were enrolled. The experimental group received orally 4 g/day of fish oil for 12 months. The primary outcome was serum TNFα levels; Secondary outcomes were IL-1β, IL-6, nitric oxide catabolites, lipoperoxides, progression on the expanded disability status scale (EDSS) and annualized relapses rate (ARR).

ELIGIBILITY:
Inclusion Criteria:

* Patients had clinically definite and magnetic resonance image supported MS
* Had at least one relapse in the year before entry into the study
* EDSS score of 0-5
* Treated with subcutaneous 250 μg interferon beta-1b (Betaseron, Bayer)

Exclusion Criteria:

* they were taking another supplement
* had progressive forms of MS
* had history of severe depression
* had history of acute liver or renal dysfunction
* had history of tobacco, drug or alcohol abuse
* had intolerance, contraindication or allergy to fish oil

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
TNF alpha | 3 months
  Serum TNF alpha levels, at baseline, 3, 6, 9 and 12 months.

SECONDARY OUTCOMES:
IL-1 beta, IL-6, Lipoperoxides, nitric oxide | 3 months
  Serum IL-1 beta, IL-6, Lipoperoxides, nitric oxide levels at baseline, 3, 6, 9 and 12 months.

OTHER OUTCOMES:
Expanded Disability Status Scale (EDSS) and Annualized rate of relapses (ARR) | 6 months
  EDSS and ARR at baseline, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Genaro G Ortiz, phD, Principal Investigator — Social Security Mexican Institute
Locations (1):
- IMSS, Specialties Hospital, Neurology Departament, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Ortiz GG, Macias-Islas MA, Pacheco-Moises FP, Cruz-Ramos JA, Sustersik S, Barba EA, Aguayo A. Oxidative stress is increased in serum from Mexican patients with relapsing-remitting multiple sclerosis. Dis Markers. 2009;26(1):35-9. doi: 10.3233/DMA-2009-0602. PMID 19242067